CLINICAL TRIAL: NCT04376385
Title: An Internet-based Self Applied Treatment Program for Prolonged Grief Disorder (PGD): A Multiple-baseline Case Series Study
Brief Title: An Internet-based Self Applied Treatment Program for Prolonged Grief Disorder (PGD)
Acronym: PGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: z7dqxrg7
Record Dates: First submitted 2020-03-23; First posted 2020-05-06 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Grief

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment condition - 9 days wait (Experimental): Internet-based Self Applied Treatment Program. Main components: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention
  Interventions: Behavioral: GROw: An Internet based Self Applied Treatment Program for Prolonged Grief Disorder (PGD)
- Treatment condition - 12 days wait (Experimental): Internet-based Self Applied Treatment Program. Main components: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention
  Interventions: Behavioral: GROw: An Internet based Self Applied Treatment Program for Prolonged Grief Disorder (PGD)
- Treatment condition - 17 days wait (Experimental): Internet-based Self Applied Treatment Program. Main components: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention
  Interventions: Behavioral: GROw: An Internet based Self Applied Treatment Program for Prolonged Grief Disorder (PGD)
- Treatment condition - 19 days wait (Experimental): Internet-based Self Applied Treatment Program. Main components: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention
  Interventions: Behavioral: GROw: An Internet based Self Applied Treatment Program for Prolonged Grief Disorder (PGD)
- Treatment condition - 33 days wait (Experimental): Internet-based Self Applied Treatment Program. Main components: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention
  Interventions: Behavioral: GROw: An Internet based Self Applied Treatment Program for Prolonged Grief Disorder (PGD)

INTERVENTIONS:
Behavioral: GROw: An Internet based Self Applied Treatment Program for Prolonged Grief Disorder (PGD) — It is a self-applied treatment through the web "psicologíaytecnología.labpsitec.es". There are 8 treatment modules. Each module lasts approximately 60 minutes. It contains written information, videos, audios, photos and interactive questionnaires. The total duration of treatment is 8-10 weeks. A support call will be made a week (maximum 10 minutes) to answer questions and reinforce and motivate the patient. No additional clinical content or counselling will be provided.
  Main components of the treatment: Motivation for change, Psychoeducation, Behavioral activation, Exposure, Mindfulness and compassion strategies, integration of loss, restoration and reconstruction of meaning, Cognitive reappraisal and Relapse prevention

SUMMARY:
The purpose os this study is examine the effect and feasibility (usability and satisfaction) of an iCBT (GROw program) for adults with PGD

DETAILED DESCRIPTION:
The death of a loved one has physical, psychological, and social consequences. Between 9.8 and 21.5% of people who lose a loved one develop Prolonged Grief Disorder (PGD). Internet- and computer-based interventions (i.e., Internet-delivered Cognitive-Behavioral Therapy, iCBT) are cost-effective and scalable alternatives that make it possible to reach more people with PGD. The main goal of the present investigation was to examine the effect and feasibility (usability and satisfaction) of an iCBT (GROw program) for adults with PGD. A secondary objective was to detect adherence to the app (Emotional Monitor) used to measure daily grief symptoms. The study had a single-case multiple-baseline AB design with six participants. The GROw program is organized sequentially in eight modules, and it is based on the dual-process model of coping with bereavement. Evaluations included a pre-to-post treatment assessment of depression, grief symptoms, and typical grief beliefs, along with daily measures of symptom frequency and intensity on the Emotional Monitor App. Treatment opinions and adherence to the App were also collected. Efficacy data were calculated using a Nonoverlap of All Pairs (NAP) analysis and Reliable Change Index (RCI).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Meeting diagnostic criterio for PGD
* Sign an informed consent
* Ability to understand and read Spanish
* Abilitiy to use a computer and having access to the Internet
* Having an e-mail address

Exclusion Criteria:

* Presence of risk of suicide or self-destructive behaviors
* Presence of another severe mental disorder (substance abuse or dependence, pshychotic disorder, dementia o bipolar disorder)
* Presence of severe personality disorder
* Presence of a medical condition whose severity or characteristics prevent the performance of treatment
* Receiving other psychological treatment during the study for PGD
* An increase and/or change in the medication during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Emotional Pain: intensity of sadness, anger, anxiety, guilt and grief | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  * Evaluation from mobile app
  Item 1: In relation to the death of your loved one; What intensity of sadness have you felt TODAY? Item2: In relation to the death of your loved one; What intensity of anger have you felt TODAY? Item 3: In relation to the death of your loved one; What intensity of anxiety have you felt TODAY? Item 4: In relation to the death of your loved one; What intensity of guilt have you felt TODAY? Item 5: In relation to the death of your loved one; What intensity of pain from loss have you felt TODAY?
  * Evaluation from mobile app

SECONDARY OUTCOMES:
Change in frequency of sad memories | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you remembered TODAY the absence of your loved one with enormous and deep sadness?
  * Evaluation from mobile app
Change in frequency of memories that produce anger | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you remembered TODAY the absence of your loved one with a huge and deep anger?
  * Evaluation from mobile app
Change in frequency of memories that produce anxiety | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you remembered TODAY the absence of your loved one with enormous and deep anxiety?
  * Evaluation from mobile app
Change in frequency of memories that produce guilt | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you remembered TODAY the absence of your loved one with a huge and deep guilt?
  * Evaluation from mobile app
Change in frequency of pleasant memories | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you had pleasant memories with your loved one TODAY?
  * Evaluation from mobile app
Change in emotion avoidance frequency | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you wished TODAY to get rid of your unpleasant emotions related to your loved one?
  * Evaluation from mobile app
Change in thoughts avoidance frequency | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you tried TODAY to get rid of unpleasant thoughts related to your loved one?
  * Evaluation from mobile app
Change in difficulty accepting the death | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you thought TODAY that you cannot believe that your beloved family has died?
  * Evaluation from mobile app
Change in difficulty accepting the death | Once a day (from the start of the baseline until the end of the treatment) and at 3 and 12 months after the end of the treatment
  Item: How often have you wished TODAY intensely that your loved one was with you?

OTHER OUTCOMES:
Satisfaction with the treatment | At the end of the treatment
  * Perceived clinical utility of each part of the treatment (0 = no useful at all; 10 = maximum utility)
  * Utility images, video, audio and written content (0 = no useful at all; 10 = maximum utility)
  * Utility, satisfaction and help in the adherence of the weekly call
Change in Prolonged Grief Disorder-13 (PG-13) | Before and after treatment, at 3 and 12 months
  Diagnostic measure. Detects prolonged grief in people who have lost a loved one. Self-administered. Duration: 10 minutes approx. Composed of 13 items. Good psychometric properties (reliability test retest Kappa coefficient = 1; Cronbach's alpha = 0.92)
Change in ADIS Clinician's severity rating scale | Before and after treatment, at 3 and 12 months
  Indicate the level of distress-interference in functioning. 1 item (from 0/"Absent" to 8/"Very severely disturbing/disabling") completed by the therapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Undecided